CLINICAL TRIAL: NCT00167817
Title: Effect of Switch to Aripiprazole on Health and Smoking Parameters in Patients With Schizophrenia: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030762
Record Dates: First submitted 2005-09-10; First posted 2005-09-14 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Smoking; Metabolic; Health; Glucose; Lipids
MeSH Terms: conditions — Schizophrenia; Smoking | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
Patients with schizophrenia are much more likely to be engaged in smoking and other addictive behaviors, possibly related to biochemical abnormalities in the reward center of the brain. The primary purpose of the present study is to investigate whether switching patients with schizophrenia to a new atypical antipsychotic, aripiprazole, a drug with a novel mechanism of action, will have an impact on smoking behavior.

DETAILED DESCRIPTION:
This is an 8 week open label trial being conducted in stable adult outpatients with schizophrenia who are smokers. The primary intervention is a switch in the subject's antipsychotic to aripiprazole, flexibly dosed between 15-30 mg/day. The outcome measures include a rating of smoking behavior using the Fagerstrom Test for Nicotine Dependence, and saliva cotinine obtained at baseline and endpoint. Secondary measures include weight, serum glucose and lipids, rating of symptom severity using the PANSS, and both ratings and instrumental measures of motor functioning. We anticipate enrolling up to 25 subjects to obtain the needed 15 completers at the week 8 endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Schizophrenia, on stable antipsychotic dose for at least one month
2. Ages 18-65 inclusive
3. Overweight (body mass index of 25 kg/m2 or greater)
4. Daily cigarette smoker (by self-report)

Exclusion Criteria:

1. Inability to provide informed consent
2. Treatment refractory schizophrenia
3. Current treatment with clozapine
4. Current antipsychotic polypharmacy which may preclude monotherapy with aripiprazole
5. Documented poor compliance with oral antipsychotic medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2003-07; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Saliva cotinine, Fagerstrom Test for Nicotine Dependence

SECONDARY OUTCOMES:
Weight
Serum glucose and lipids
Rating of symptom severity using the PANSS
Ratings and instrumental measures of motor functioning

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Meyer, MD, Principal Investigator — University of California, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States